CLINICAL TRIAL: NCT00991744
Title: Phase III Randomised Study on Liposomal Cytarabine (DepoCyte®) vs. Intrathecal Triple for CNS-Treatment During Maintenance Therapy in High-Risk Acute Lymphoblastic Leukemia Patients in NOPHO ALL 2008 Treatment Protocol
Brief Title: Liposomal Cytarabine for Central Nervous System (CNS)-Treatment in High-risk Acute Lymphoblastic Leukemia (ALL)
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Sterility problems in DepoCyte production
Sponsor: Nordic Society for Pediatric Hematology and Oncology (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Arja Harila-Saari, Associate professor, Nordic Society for Pediatric Hematology and Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOPHOALL2008-DepoCyte
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Leukemia; Central nervous system; Neurotoxicity; Liposomal cytarabine; Children; Acute lymphoblastic leukemia; Childhood acute lymphoblastic leukemia; Intrathecal; Efficacy; Safety
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Neurotoxicity Syndromes | interventions — Cytarabine; Methylprednisolone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal cytarabine (Experimental): Intrathecal liposomal cytarabine (25 - 50 mg) combined with intrathecal prednisolone sodium succinate and oral dexamethasone 6 times during maintenance treatment for high-risk ALL
  Interventions: Drug: Liposomal cytarabine
- Intrathecal triple (Active Comparator): Intrathecal methotrexate, cytarabine and prednisolone
  Interventions: Drug: Intrathecal triple

INTERVENTIONS:
Drug: Liposomal cytarabine — Intrathecal liposomal cytarabine combined with intrathecal prednisolone and oral dexamethasone during maintenance treatment for high-risk ALL
  Other Names: Cytarbine; Ara-C; Cytosar-U; Cytosine arabinoside; Precortalon; Di-Adreson F
  Arms: Liposomal cytarabine
Drug: Intrathecal triple — Intrathecal methotrexate (8-12 mg), cytarabine (20 - 30 mg) and prednisolone sodium succinate (12,5 - 20 mg) 6 times during maintenance treatment in high-risk ALL protocol
  Other Names: DepoCyte; DepoCyt; Precortalon; Di-Adreson-F; Cytarabine; Ara-C; Cytosar-U; Cytosine arabinoside
  Arms: Intrathecal triple

SUMMARY:
* Replacement of intrathecal Triple (methotrexate, cytarabine, prednisolone) with intrathecal liposomal cytarabine and prednisolone during maintenance therapy will decrease the CNS relapse rate in high-risk ALL patients.
* Both acute and long-term toxicity are equal in both treatment arms.

DETAILED DESCRIPTION:
20% of children with ALL still fails to be cured. The ALL-2008 protocol is a treatment and research protocol that aims to improve the overall outcome of Nordic children and adolescents with ALL in comparison with the ALL-2000 protocol and previous NOPHO protocols.

The specific and primary objectives of the randomised study is:

1. To replace intrathecal triple (methotrexate, cytarabine and glucocorticosteroid) by intrathecal liposomal cytarabine and glucocorticosteroid during maintenance therapy in order to decrease the central nervous system relapse rate in high-risk acute lymphoblastic leukemia patients.
2. To evaluate acute and long-term toxicity in both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* High risk acute lymphoblastic leukemia
* Not eligible for bone marrow transplantation
* Age 1-18
* Written informed consent has been obtained

Exclusion Criteria:

* Persistent NCI grade 3-4 neurotoxicity from previous treatments
* Bilineage ALL
* Leukemia predisposing syndromes (e.g. Downs syndrome, Ataxia Telangiectasia)
* Previous cancer
* Known intolerance to NOPHO ALL 2008 anticancer agents
* Sexually active females will use safe contraceptives
* Previous treatment with intrathecal liposomal cytarabine

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of leukemia relapses in the central nervous system | 5 years

SECONDARY OUTCOMES:
Neurological toxicity | 6 months after cessation of leukemia therapy

CONTACTS AND LOCATIONS:
Overall Officials: Arja Harila-Saari, MD, Principal Investigator — Oulu University Hospital
Locations (5):
- Department of Pediatrics, Rigshospitalet, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- University of Reykjavik, Iceland, Reykjavik, Iceland
- University Hospital of Trondheim, Norway, Trondheim, Norway
- Department of Pediatrics, Drottning Sylvias Pediatric Hospital, Gothenburg, Sweden